CLINICAL TRIAL: NCT03909516
Title: A Post-Market, Prospective Study to Evaluate the Iovera° Device in Treating Pain Associated With Anterior Cruciate Ligament Reconstruction
Brief Title: Evaluate the Iovera° Device in Treating Pain Associated With Anterior Cruciate Ligament Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Myoscience recently acquired - decided to redesign study.
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYO-1378
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-04

CONDITIONS: ACL Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Adductor Canal Block required, the formulation, or "cocktail," of medications used are to be recorded in the medical record. Start and end time will be recorded.
- Standard of Care + iovera° Treatment (Active Comparator): The iovera° device will be prepared by the trained Anesthesiologist User Guide. If at any time the device does not perform as expected the Investigator and Anesthesiologist will follow procedures as outlined in the User Guide. Start and end time will be recorded.
  Once localized anesthesia of the block area is achieved, the Anesthesiolgist, or designee, will complete the iovera° treatment. Upon completion of block, The Anesthesiologist or designee will assess the treatment areas for adverse events.
  Adductor Canal Block required, the formulation, or "cocktail," of medications used are to be recorded in the medical record. Start and end time will be recorded.
  Local Infiltration Analgesia - 20cc 0.5% ropivicaine only
  Interventions: Device: iovera°

INTERVENTIONS:
Device: iovera° — The iovera° device will be prepared by the trained Anesthesiologist User Guide. If at any time the device does not perform as expected the Investigator and Anesthesiologist will follow procedures as outlined in the User Guide. Start and end time will be recorded. Once localized anesthesia of the block area is achieved, the Anesthesiolgist, or designee, will complete the iovera° treatment. Upon completion of block, The Anesthesiologist or designee will assess the treatment areas for adverse events. Adductor Canal Block required, the formulation, or "cocktail," of medications used are to be recorded in the medical record. Start and end time will be recorded.
  Local Infiltration Analgesia - 20cc 0.5% ropivicaine only
  Arms: Standard of Care + iovera° Treatment

SUMMARY:
To evaluate the outcomes of patients undergoing iovera° treatment of the ISN, AFCN and LFCN on postoperative knee pain and function following anterior cruciate ligament reconstruction

DETAILED DESCRIPTION:
The most commonly reconstructed ligament in the knee is the anterior cruciate ligament (ACL). In 2006 a total of 134,421 ACL reconstructions were performed in the United States, representing a 37% increase in procedures since 19941. Today, most ACL reconstructions are performed on an outpatient basis. While this has led to improvements in patient satisfaction and cost, it has simultaneously resulted in more complicated postoperative pain management. Managing this pain via multi-modal strategies, including peripheral nerve blocks, in the postoperative phase has been shown to decrease opioid related side effects, decrease hospital stay, and increase time to ambulation. Nursing, hospital, and pharmacy utilization in managing PCA, continuous regional nerve blocks, and administration of oral opioid dosing are associated with higher costs of care and introduce sources for staff error. Furthermore, the idea of multi-modal pain management extends beyond the surgical procedure. Decreasing prescription opioid use during outpatient rehabilitation decreases NSAID and opioid related side effects.

Myoscience, Inc. (Fremont, CA) has developed a device - iovera° - as a novel, minimally-invasive procedure using cold to target sensory nerve tissue and provide temporary pain relief through cryoneurolysis. The iovera° device uses well-established principles of cryobiology to temporarily deactivate sensory nerves that contribute to pain. Prior studies of the iovera° device have provided evidence of effectiveness and safety for treatment of the Infrapatellar Branch of the Saphenous Nerve and another study has demonstrated that a short-term block of this nerve resulted in reduced pain following an ACL reconstruction.

In a multicenter, double-blind, sham-controlled, randomized trial sponsored by Myoscience, Inc, the iovera° device was shown to temporarily relieve pain in patients with osteoarthritis of the knee. Compared to the sham group, patients who received active treatment had a statistically significant greater change from baseline in the WOMAC pain subscale score at Day 30 (p=0.0004), Day 60 (p=0.0176), and Day 90 (p=0.0061). Patients deemed WOMAC pain responders at Day 120 continued to experience a statistically significant treatment effect at Day 150. Most expected side effects were mild in severity and resolved within 30 days. The incidence of device- or procedure-related adverse events was similar in the two treatment groups with no occurrence of serious or unanticipated adverse events.

The goal of the study described herein is to determine the safety and efficacy of the iovera° treatment for reducing the pain associated with anterior cruciate ligament (ACL) reconstruction

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age
2. Scheduled to undergo unilateral anterior cruciate ligament reconstruction with patellar tendon autograft quadricep tendon autograft or hamstring tendon autograft
3. In the opinion of the investigator, the subject is an active participant in recreational or competitive sports, physical activity, or other fitness regimen at the time of ACL injury and is seeking reconstruction to help return to sport or activity
4. Subject is willing and able to give written informed consent.
5. Subject is fluent in verbal and written English.
6. Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
7. Subject is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the Investigator's opinion, exposes the Subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Chronic opioid use (defined as daily or almost daily use of opioids for >3 months).
2. Prior ligamentous injury and/or surgery of the operative knee (arthroscopic surgeries allowed) or relevant musculoskeletal impairment
3. Prior surgery or injury in the knee or treatment areas that may have altered the anatomy of the target nerves or resulted in scar tissue in the iovera° treatment areas.
4. Any pain disorder, neuro-muscular disorder, or neuropathy that in the opinion of the Investigator may confound post-operative assessments for pain or rehabilitation. Examples include but are not limited to: fibromyalgia, diabetic neuropathy, multiple sclerosis, etc.
5. History of opioid or alcohol abuse within past 3 years and/or active opioid user for other medical conditions.
6. Open and/or infected wound in the treatment areas or any local skin condition at the treatment sites that in the Investigator's opinion would adversely affect treatment or outcomes.
7. History of cryoglobulinemia
8. History of paroxysmal cold hemoglobinuria.
9. History of cold urticaria.
10. History of Raynaud's disease.
11. Any chronic medical condition that in the Investigator's opinion would prevent adequate participation.
12. Any chronic medication use (prescription, over-the-counter, etc.) that in the Investigator's opinion would affect study participation or Subject safety.
13. For any reason, in the opinion of the Investigator, the Subject may not be a suitable candidate for study participation (i.e., worker's compensation, history of noncompliance, drug dependency, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Average Daily Pain (ADP) Intensity Scores | Baseline to 10 days post-surgery
  The primary endpoint is the change from baseline to 10 days post-surgery in mean Average Daily Pain (ADP) Intensity Scores for iovera patients compared to standard of care.
  Trial success is demonstrated under the primary hypothesis if the p-value corresponding to the study t-test for the effect of iovera compared to the standard of care group from baseline is less than or equal to 0.05.
Pill Count | Baseline to 12 Week
  Amount of pills taken - medications to be recorded include prescription opioids. The investigator, or their designee, will then count the number of pills remaining in the bottle, record this amount and return the pills to the Subject.

SECONDARY OUTCOMES:
Area-Under-Effect (AUE) curves | Baseline to 12 Week
  Area-Under-Effect (AUE) curves of the change in ADP-intensity scores
Single Assessment Numerical Evaluation (SANE) Score | Baseline to 12 Week
  The Single Assessment Numerical Evaluation (SANE) score was introduced as a tool to aid in the assessment of clinical outcomes by decreasing the burden of gathering outcomes data without limiting the meaningfulness of the data. It has been demonstrated to be a reliable reflection of knee symptoms after anterior cruciate ligament (ACL) reconstruction in both male and female subjects. The SANE score has been subjected to rigorous statistical evaluation and has proven to be a valid and responsive patient-reported outcome measure. The SANE score is determine by the subject's response to the following question:
  "On a scale of 0 to 100, how would you rate your knee's function, with 100 being normal?"
Knee Injury and Osteoarthritis Outcomes Score (KOOS JR.) | Baseline to 12 Week
  The KOOS JR. score consists of 7 questions from 3 subscales: Stiffness (1 question), Pain (4 questions), and Function in daily living (2 questions). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from None (0) to Extreme (4). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated. A copy of the KOOS JR. is located in Attachment 1. After completion by the Subject, the study coordinator or designee will enter the data into the CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rivadeneyra, MD, Principal Investigator — HOAG

IPD SHARING:
Plan to Share IPD: No